CLINICAL TRIAL: NCT03809572
Title: Mechanisms of Action of MBCT-PD: A Pilot Study
Brief Title: Mindfulness Based Cognitive Therapy (MBCT) During Pregnancy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to restrictions to in-person research due to COVID-19
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kristen Mackiewicz Seghete, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1R21AT010292-01 (NIH)
Record Dates: First submitted 2019-01-11; First posted 2019-01-18 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Maternal Psychological Distress; Postpartum Depression; Prenatal Stress
Keywords: fMRI; pregnancy; postpartum; MBCT; Mindfulness Based Cognitive Therapy; emotion regulation
MeSH Terms: conditions — Depression, Postpartum; Emotional Regulation | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: The study is a randomized, control trial with an intervention arm, Mindfulness Based Cognitive Therapy (MBCT) adapted for pregnant women (Dimidjian, Goodman, et al., 2016), and treatment as usual (TAU) arm. The study will be blinded to staff (except for the study coordinator(s) and interventionists), but participant blinding is not possible due to the nature of the intervention. Participants will be randomized using a stratified block design after initial eligibility determination. Randomization will be stratified based on current depressive symptoms and current stress levels.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Given the use of group therapy, participants and interventionists cannot be blinded to group assignment. The study is designed to minimize the extent to which study staff, aside from interventionists and the primary Study Coordinator(s), are aware of group assignment. The Study Coordinator(s) needs to know group assignment because they will inform participants of their group assignment and will be the main point of contact for participants throughout the study, as to reduce risk of participants revealing their group assignment to other study staff. Participants will be informed that only the Study Coordinator(s) and interventionists, if applicable, are aware of their group assignment. Therefore, in order to ensure the integrity of the research study, they should refrain from discussing their group assignment with other staff members.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Cognitive Therapy (Experimental): Mindfulness Based Cognitive Therapy (MBCT) adapted for pregnancy includes 8 sequential, weekly 2-hour group sessions co-led by two master's level therapists. Sessions include: 1) introducing new mindfulness skills through in-session practice, 2) reviewing mindfulness practices and troubleshooting barriers to practice, 3) reinforcing mindfulness skills through in-session practice and debriefing, 4) learning about how thoughts influence feelings and behaviors (not all sessions), 5) providing psychoeducational information to support skills, and 6) encouraging the establishment of social support.
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy
- Treatment as usual (TAU) (No Intervention): All participants will receive routine prenatal care from an identified medical provider, which they have initiated on their own. They will be able to engage in any services recommended by their primary medical provider or that they voluntarily initiate. For ethical reasons, they are not prohibited from engaging in any type of therapeutic, complementary, or medication treatment (after enrollment). The TAU group will be offered a delayed treatment option, after the 6 month follow-up. This will be a 2 hour mindfulness psychoeducation session, offered between 6 and 9 months postpartum. Several core mindfulness concepts included in the full MBCT curriculum will be taught and participants will complete several brief mindfulness activities.

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — See Arm description
  Other Names: Mindfulness Based Cognitive Therapy for Perinatal Depression
  Arms: Mindfulness Based Cognitive Therapy

SUMMARY:
The study is a pilot randomized control trial of a validated intervention, Mindfulness Based Cognitive Therapy (MBCT) adapted for pregnancy, developed to reduce risk for postpartum depression. This study examines emotion regulation as a potential mechanism of action, at both the behavioral and neurobiological level, that carries forward to the postpartum period. A secondary mechanism of action to be explored is cognitive control. This study will also consider other potential influences on treatment response and psychiatric outcomes, including perinatal stress and depressive symptoms. The study population is pregnant women age 21-45.

DETAILED DESCRIPTION:
The study will involve an online screen of potentially eligible pregnant women. If participants are eligible after the online screen, they will be invited in for an in person assessment, including cognitive testing and a diagnostic interview, to determine eligibility. After the assessment, they will be informed of their eligibility status and, if applicable, randomized to Mindfulness Based Cognitive Therapy (MBCT) or treatment as usual (TAU). Participants in the MBCT group will complete 8 weekly, 2 hr group therapy sessions during pregnancy, as well as receive TAU. The TAU group will engage in regular care during pregnancy and be offered the option to attend one mindfulness psychoeducation session postpartum. Participants in the MBCT group will complete questionnaires prior to the 1st group session, after the 4th session, and after the 8th/final session. Participants in the TAU group will complete the same questionnaires at equivalent time points. All participants will come in for an in-person session at 34 weeks GA, during which they will complete questionnaires and a brief clinical interview. Participants will come in for an MRI scan session at 6 weeks postpartum. In addition to structural and functional MRI scanning, they will also complete questionnaires, a cognitive task, and brief psychiatric interview. At 6 months postpartum, participants will return for a visit, during which they will complete questionnaires, cognitive measures, and a clinical interview. This will be the final visit for women in the MBCT group. Women in the TAU group will complete a singe mindfulness psychoeducation session between 6 and 9 months postpartum; this must occur after their 6 month visit. Some visits will be adapted as needed to accommodate institutional requirements with regard to restrictions due to COVID-19.

ELIGIBILITY:
Inclusion:

1. female who is currently pregnant (8-22 weeks gestational age (GA) at time of screen)
2. 21-45 years old
3. single gestation
4. fluently speak English
5. be available and physically able to attend scheduled group meetings
6. have a prior history of at least 1 major depressive episode (as determined through psychiatric interviewing).

Exclusion (at enrollment):

1. Magnetic Resonance Imaging (MRI) contraindication (e.g., metal in their body)
2. major neurological or medical illness (e.g., diabetes, multiple sclerosis)
3. history of head trauma (loss of conscious > 2 minutes)
4. Intelligence Quotient (IQ) < 80
5. uncorrectable vision or hearing impairments (including color blindness)
6. use of psychotropic medications, corticosteroids, insulin, or any other medications that might impact the central nervous system
7. current illicit drug use or diagnosis of a current substance use disorder
8. current diagnosis of an eating disorder
9. current depressive or manic episode
10. diagnosis of a neurodevelopmental disorder (Autism, Intellectual Disability)
11. any history of psychosis
12. current active suicidality and/or homicidality, or interpersonal violence
13. prior history of engaging in mindfulness-based psychotherapeutic interventions (e.g., Mindfulness Based Cognitive Therapy (MBCT), Mindfulness Based Stress Reduction (MBSR), Dialectical Behavior Therapy (DBT))
14. known congenital, genetic, or neurologic disorder of the fetus (e.g., Down syndrome, fragile X)
15. pregnancy-specific medical conditions or complications that significantly increase risk (e.g., placental separation, placenta previa)
16. History of meningitis or seizures (except infantile or febrile)

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale - Revised (CESD-R) | 6 Weeks Postpartum
  Self-reported depressive symptoms over the past two weeks. There are 20 items, each scored from 0-4. The total score range is from 0-80. Total score will be used, with higher scores indicate more depressive symptoms.
Emotion Regulation Questionnaire (ERQ) | 6 Weeks Postpartum
  Self-report of emotion regulation skills. There are two primary subscales, cognitive reappraisal (range: 6-42) and expressive suppression (range: 4-28). Outcome will be total score on the cognitive reappraisal scale. Higher scores for reappraisal indicate better emotion regulation.
Stroop Task | 6 Weeks Postpartum
  The classic Stroop task is a robust measure of cognitive control. Participants will view a color word in a different color ink, naming the ink color. A control condition is included with neutral words. Interference score will be calculated using reaction times.
Brain activation during an emotion regulation task | 6 Weeks Postpartum
  An emotion regulation task will be completed during a functional magnetic resonance imaging (fMRI) scan in order to examine whole-brain functional activation. Individuals will view negative and neutral pictures from the International Affective Picture System. For some pictures, they will just view the images. For some negative pictures, they will be asked to regulate their responding using a distancing technique that has been introduced to them.
Brain activation during the Stroop task | 6 Weeks Postpartum
  The Stroop task will be completed during a functional magnetic resonance imaging (fMRI) scan in order to examine whole-brain functional activation when cognitive control must be exerted.

SECONDARY OUTCOMES:
Rate of Postpartum Depression | 6 Weeks Postpartum, 6 Months Postpartum
  Presence of a major depressive episode will be used to determine the presence of postpartum depression. Major depressive episodes will be assessed using the Mood Module of the Structured Clinical Interview for the Diagnostic and Statistical Manual, Fifth Edition (SCID-5).
Emotion Regulation Questionnaire (ERQ) | 6 Months Postpartum
  Self-report of emotion regulation skills. There are two primary subscales, cognitive reappraisal (range: 6-42) and expressive suppression (range: 4-28). Outcome will be total score on the cognitive reappraisal scale. Higher scores for reappraisal indicate better emotion regulation.
Stroop Task | 6 Months Postpartum
  The classic Stroop task is a robust measure of cognitive control. Participants will view a color word in a different color ink, naming the ink color. A control condition is included with neutral words. Interference score will be calculated using reaction times.
Infant Behavior Questionnaire - Revised (IBQ-R) | 6 Months Postpartum
  A 193 item self-report measure completed by mothers about specific temperament-related behaviors displayed by their infant over the past two weeks. There are 14 sub-scales derived, each ranging from 0-7. A negative emotionality composite will be derived from the fear, sadness, and distress to limitations sub-scales.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Mackiewicz Seghete, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
We propose to share de-identified individual participant data that underlie the results of this study, with proper approval.
Supporting Information: Study Protocol, SAP
Time Frame: 12 months after final data collection is concluded through 5 years after publication
Access Criteria: The Principal Investigator (PI) will review requests for individual participant data (IPD). IPD will be provided with appropriate Institutional Review Board (IRB) approval or determination of IRB exemption and approval by the National Center for Complementary and Integrative Health (NCCIH) program officer. IPD may be provided to investigators associated with a university or reputable research institution with an associated IRB. De-identified IPD will be provided through a secure sharing mechanism.

REFERENCES:
- [Background] Dimidjian S, Goodman SH, Felder JN, Gallop R, Brown AP, Beck A. Staying well during pregnancy and the postpartum: A pilot randomized trial of mindfulness-based cognitive therapy for the prevention of depressive relapse/recurrence. J Consult Clin Psychol. 2016 Feb;84(2):134-45. doi: 10.1037/ccp0000068. Epub 2015 Dec 14. PMID 26654212